CLINICAL TRIAL: NCT06625333
Title: A Prospective Non-interventional Study to Evaluate Clinical Outcomes of Ribociclib Combined With Endocrine Therapy in Elderly Patients With HR+HER2 - Advanced Breast Cancer in Routine Clinical Practice in Russian Federation
Acronym: PARFENOPA
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ARU06
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HR+HER2- Advanced Breast Cancer
Keywords: HR+HER2- advanced breast cancer, ribociclib, elderly patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is а prospective, non-interventional, primary data collection study to evaluate the effectiveness, safety and quality of life in older patients (≥65 years) with HR+HER2- advanced breast cancer receiving ribociclib with ET in the first or second line in the real-life settings in Russia.

DETAILED DESCRIPTION:
In this study, an index event is a start of ribociclib+ET treatment. Post-index follow-up period is 24 months or until treatment discontinuation. The recruitment period is planned for 12 months. The interim analyses will be performed after enrollment is complete, and further one year later. Patients will visit the sites in accordance with routine clinical practice. It is assumed according to the clinical practice that visits will be conducted every 3-4 months. Patients will undergo standard procedures and tests according to clinical guidelines and physician's judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years at the moment of ribociclib+ET initiation
2. Female/Male gender
3. Confirmed diagnosis of locally advanced/metastatic not eligible for curative surgery HR+HER2- BC for whom the treating physician took the decision to initiate treatment with ribociclib+IA/FUL in the first or in the second line of the treatment
4. Patient who initiated treatment with ribociclib+IA/FUL no longer than 4 weeks (28 days) prior to written informed consent for this study
5. Provision of written informed consent.

Exclusion Criteria:

1. Patients with a life expectancy of less than 3 months per the investigator's judgment
2. Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. (Patients participating in other investigator initiated research or NIS can be included as long as their standard of care is not altered by the study)
3. Patients on active treatment for malignancies other than aBC within 3 years before BC diagnosis
4. Patients with active cardiac disease, or history of cardiac dysfunction, including prolonged QT interval corrected using Fridericia's formula (QTcF > 450 msec).

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients with HR+HER2- advanced breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
change of QoL (RAND SF-36) | from baseline to the level at 12 months
  The primary endpoint of the study is the change of QoL during treatment with ribociclib+ET from baseline to the level at 12 months (RAND SF-36) across all age's subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) and depend on treatment lines (first-line (1L) or in second-line (2L) settings)

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | up to two years
  Time to treatment failure (TTF) in HR+/HER2- aBC women initiating treatment with ribociclib+ET across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L)
Progression free survival rate (PFS) | up to two years
  Progression free survival rate (PFS) at 24 months in HR+/HER2- aBC women initiating treatment with ribociclib+ET across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L)
Median progression free survival | up tp two years
  Median progression free survival (if reached) in HR+/HER2- aBC women initiating treatment with ribociclib+ET across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L)
Overall survival rate (OS) | up to two years
  Overall survival rate (OS) at 24 months in HR+/HER2- aBC women initiating treatment with ribociclib+ET in across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L)
Objective response rate (ORR) | up to two years
  Objective response rate (ORR) as assessed by the investigator in HR+/HER2- aBC women initiating treatment with ribociclib+ET across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L)
Clinical benefit rate (CBR) | up to two years
  Clinical benefit rate (CBR) as assessed by the investigator in HR+/HER2- aBC women initiating treatment with ribociclib+ET across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) depend on treatment lines (1L or 2L).
Proportions (%) of patients and reasons of permanent discontinuation of ribociclib | up to two years
  Proportions (%) of patients and reasons of permanent discontinuation of ribociclib
Proportions (%) of patients and reasons of dose adjustment on ribocicli | up to two years
  Proportions (%) of patients and reasons of dose adjustment on ribocicli
Adverse events (AEs) frequency and severity | up to two years
  Adverse events (AEs) frequency and severity
Quality of life (RAND SF-36, questionnaire of patient's satisfaction) | up to two years
  Quality of life (RAND SF-36, questionnaire of patient's satisfaction) during treatment with ribociclib + ET (AI/FUL) across all age subgroups (ages 65 to 74 years; middle-old, 75 to 84 years; and oldest-old, ≥85 years) and in first-line (1L) and in second-line (2L) settings

CONTACTS AND LOCATIONS:
Locations (19):
- Russia (19):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Bryansk
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Khabarovsk
  - Novartis Investigative Site, Khanty-Mansiysk
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tambov
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No